CLINICAL TRIAL: NCT06251063
Title: Improving Social Relationships for Adolescents with Central Disorders of Hypersomnolence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Eric Zhou, PhD, Assistant Professor, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00047080
Record Dates: First submitted 2024-01-23; First posted 2024-02-09 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Narcolepsy Type 1; Narcolepsy Type 2; Idiopathic Hypersomnia
Keywords: Narcolepsy Type 1; Narcolepsy Type 2; Central Disorders of Hypersomnolence; Idiopathic Hypersomnia; Social Relationships; Adolescents
MeSH Terms: conditions — Idiopathic Hypersomnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Web-based psychoeducational Resource (Experimental): Eligible families will be provided with website access instructions. Parents and children will be instructed to review the materials separately. The intervention will provide each person with individualized action items to be discussed as a family. It is anticipated that reviewing all of the psychoeducational materials will take the parent/child approximately one hour, resulting in a total intervention burden of two hours for the family. Participants will be encouraged to return to the website as often as needed to review content. For the purposes of this project, they will be instructed to review all intervention materials within one month of receiving the website access instructions.
  Interventions: Behavioral: Web-based psychoeducational resource

INTERVENTIONS:
Behavioral: Web-based psychoeducational resource — The website will incorporate animations/illustrations to enhance comprehension, patient stories, and video-based expert explanations.
  The materials will address the following content areas:
  * Provide families with data demonstrating how prevalent social relationship struggles are for children with CDH.
  * Describe specific social challenges that commonly affect children with CDH.
  * Explain the impact that medications typically prescribed for CDH may have on social relationship health.
  * Help families advocate for their child's social needs at school.
  * Support children and their families in decision-making about appropriate disclosure with peers at school and in extracurricular settings.
  * Offer strategies to support families in raising the issue of social relationship health with the child's sleep physician.
  * Provide a list of programming which offers children both structured and unstructured opportunities for social engagement

SUMMARY:
The goal of this study is to test a web-based psychoeducational resource for adolescents with central disorders of hypersomnolence and their families. The investigators hope to assess the website's usability, acceptability, and feasibility, as well as its potential effect on social relationship health.

Participants will be asked to review the content of the psychoeducational websites. The participants will then provide feedback on the website, as well as the adolescent's social relationships and social health before and after reviewing the website through online surveys.

DETAILED DESCRIPTION:
The American Academy of Sleep Medicine's clinical practice guideline task force concluded that "reliance on medications alone to treat CNS hypersomnia conditions is likely insufficient." Our stakeholder data demonstrated that this issue is a significant challenge in the domain of social relationship health for children with narcolepsy type 1 and 2 (NT1/NT2) and idiopathic hypersomnia (IH). With one peak for symptom onset in adolescence, a critical period in a child's social development, children with NT1/NT2/IH and their families report significant social sequelae of the disorder and its treatment that have lifelong implications. To address this important, yet consistently overlooked real-life concern for adolescents with CDH, the investigators intend to assess an online psychoeducational website that the investigators designed to provide families with the knowledge and resources to improve the adolescent's social relationship health.

A total of 45 families will participate in a single-arm usability, feasibility, and acceptability trial. Eligible families will be provided with instructions on how to access the website. Participants will be encouraged to return to the website as often as needed to review content. For the purposes of this study, participants will be instructed to review all intervention materials within one month of receiving website access. The participants will then complete feedback questionnaires on the secure online platform REDCap. This study will inform a future randomized controlled trial testing the efficacy of the investigators' intervention. The investigators' stakeholder informed program will be the first of its kind for children with NT1/NT2/IH, with the potential to be widely disseminated.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent from 10-17 years of age and parent of the adolescent
* Adolescent has physician-diagnosed narcolepsy type 1 or type 2, or idiopathic hypersomnia
* English fluency
* Interest in learning more about how to improve social health for adolescents with a CDH

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Usability | 5 weeks
  System Usability Scale. The minimum score is 10 and the maximum score is 50. Each question is measured on a scale from 1-5. A higher score indicates higher usability (better outcome). Completed by both the parent and child.
Acceptability (Enrollment) | 5 weeks
  Proportion of eligible families who express interest in the study choosing to enroll.
Acceptability (Satisfaction) | 5 weeks
  Satisfaction subscale of the Usability, Satisfaction, and Ease of use scale. Each question is measured on a scale from 1-7. The minimum score is 7 and the maximum score is 49. A higher score indicates higher website satisfaction (better outcome).
Acceptability (Recommend Website) | 5 weeks
  Proportion of participants who respond positively to the Post-Intervention questionnaire item "Would you recommend this website to other families of children with NT1/NT2/IH?".
Feasibility (Website Access) | 5 weeks
  Proportion of participants that access the website at least once during the study period.
Feasibility (Assessment Completion) | 5 weeks
  Proportion of participants who complete the Post-Intervention Assessment.

SECONDARY OUTCOMES:
Relationship Quality | 0 weeks and 5 weeks
  Patient Reported Outcomes Measurement Information System Pediatric Peer Relationships Scale (PROMIS-PPRS). Each question is measured on a scale of 0-4. The minimum score is 0 and the maximum score is 32. A higher score means better peer relationships (better outcome).
Social Problems (Loneliness) | 0 weeks and 5 weeks
  UCLA Three-Item Loneliness Scale. Completed by patient and parent. Each question is measured on a scale of 1-3. The minimum score is 3 and the maximum score is 9. A higher score means more loneliness (worse outcome).
Social Problems (Social Relationships) | 0 weeks and 5 weeks
  NIH Toolbox Pediatric Social Relationship Scales. Using the Emotional Support, Friendship, and Perceived Rejection Items. Each question is measured on a scale of 1-5. The minimum score is 19 and the maximum score is 95. A higher score means better social relationships (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Zhou, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou ES, Revette A, Heckler GK, Worhach J, Maski K, Owens JA. Building a deeper understanding of social relationship health in adolescents with narcolepsy disorder. J Clin Sleep Med. 2023 Mar 1;19(3):491-498. doi: 10.5664/jcsm.10372. PMID 36468655